CLINICAL TRIAL: NCT01725282
Title: Phase 2 Study of FK949E - Double-blind, Placebo-controlled, Comparative Study in Major Depressive Disorder Patients With Inadequate Response to Existing Antidepressants
Brief Title: Study to Evaluate the Effect and Safety of Quetiapine Extended Release (XR) (FK949E) in Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6949-CL-0005
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder
Keywords: patients; FK949E
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received matching placebo tablets once daily before bedtime for 7 weeks.
  Interventions: Drug: Placebo
- Quetiapine 50 mg (Experimental): Participants received quetiapine extended release (XR) 50 mg tablets once daily before bedtime for 7 weeks.
  Interventions: Drug: quetiapine extended release (XR)
- Quetiapine 150 mg (Experimental): After 2 days of up-titration, participants received quetiapine XR 150 mg tablets once daily before bedtime for 6 weeks followed by quetiapine XR 50 mg tablets once daily for 1 week.
  Interventions: Drug: quetiapine extended release (XR)
- Quetiapine 300 mg (Experimental): After 4 days of up-titration, participants received quetiapine XR 300 mg tablets once daily before bedtime for 6 weeks followed by quetiapine XR 150 mg tablets once daily for 1 week.
  Interventions: Drug: quetiapine extended release (XR)

INTERVENTIONS:
Drug: quetiapine extended release (XR) — Extended release tablets
  Other Names: Seroquel XR; FK949E
  Arms: Quetiapine 150 mg; Quetiapine 300 mg; Quetiapine 50 mg
Drug: Placebo — matching tablets
  Arms: Placebo

SUMMARY:
In this study, quetiapine XR or placebo will be administered orally for 6 weeks to major depressive disorder patients with lack of response to existing antidepressants, with the aim of evaluating the efficacy of quetiapine XR and dose-response in three quetiapine XR dose groups based on changes in Montgomery-Asberg Depression Rating Scale (MADRS) scores.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder as specified in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR) with the use of the Mini-International Neuropsychiatric Interview (M.I.N.I.)
* Documented appropriate treatment history (i.e., lack of response to treatment at labeled dosage for at least 4 weeks) for the current major depression episode with an antidepressant other than that used concomitantly with the study drug
* The Hamilton Depression Rating Scale (HAM-D17) total score of 20 points or more and HAM-D17 depressed mood score of 2 points or more

Exclusion Criteria:

* Concurrent or previous history of DSM-IV-TR Axis I disorders, except major depressive disorder, within the last 6 months before informed consent
* Concurrence of DSM-IV-TR Axis II disorder that is considered to greatly affect patient's current mental status
* The duration of the current major depression episode is shorter than 4 weeks or longer than 24 months at informed consent
* History of dependence of substances other than caffeine and nicotine or history of abuse or dependence of alcohol
* The HAM-D17 suicide score of 3 points or more, history of suicide attempt within the last 6 months before informed consent, or the risk of suicide in the investigator's or subinvestigator's opinion
* Concurrent or previous history of diabetes mellitus. HbA1c levels of 6.1% (Japan Diabetes Society values) or more within the past 2 months
* Electroconvulsive therapy within the last 62 days before primary registration (within the last 90 days before secondary registration)
* Treatment with a depot antipsychotic within the last 28 days
* Documented or suspected (to be a carrier of) conditions such as renal failure, hepatic failure, serious cardiac disease (or current use of antiarrhythmic drugs), hepatitis B, hepatitis C, or acquired immunodeficiency syndrome (AIDS)
* Concurrence of uncontrolled hypertension (defined as a systolic blood pressure of 180 mmHg or more, or a diastolic blood pressure of 110 mmHg or more at primary registration) or unstable angina that may worsen with the study or may affect the study results based on the clinical judgment of the investigator or subinvestigator
* Concurrence of hypotension (defined as a systolic blood pressure of less than 100 mmHg at primary registration) or orthostatic hypotension
* Concurrence of malabsorption syndrome, hepatic disease, or other conditions that may affect the absorption and/or metabolism of the study drug
* Concurrent or previous history of cerebrovascular disease or transient ischemic attack (TIA)
* Known hypersensitivity to quetiapine or any component of FK949E tablets

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2011-12-14 (Actual); Primary Completion 2013-08-24 (Actual); Study Completion 2013-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (3):
- Japan (3):
  - Hokkaidou
  - Kantou
  - Kinki

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Fukushi R, Nomura Y, Katashima M, Komatsu K, Sato Y, Takada A. Approach to Evaluating QT Prolongation of Quetiapine Fumarate in Late Stage of Clinical Development Using Concentration-QTc Modeling and Simulation in Japanese Patients With Bipolar Disorder. Clin Ther. 2020 Aug;42(8):1483-1493.e1. doi: 10.1016/j.clinthera.2020.06.002. Epub 2020 Aug 11. PMID 32792252
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=180

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Quetiapine 50 mg | Quetiapine 150 mg | Quetiapine 300 mg
Started | 44 | 44 | 41 | 43
Completed | 42 | 39 | 33 | 36
Not Completed | 2 | 5 | 8 | 7
Not completed — Adverse Event | 1 | 3 | 6 | 4
Not completed — Exacerbation of Target Disease | 1 | 0 | 0 | 1
Not completed — Met Exclusion Criteria | 0 | 0 | 1 | 0
Not completed — Study Site Withdrawal | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Quetiapine 50 mg | Quetiapine 150 mg | Quetiapine 300 mg | Total
Number analyzed (Participants) | 44 | 44 | 41 | 43 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (11.2) | 39.0 (9.5) | 35.2 (8.6) | 37.3 (9.7) | 37.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 17 | 17 | 68
  Male | 25 | 29 | 24 | 26 | 104
Region of Enrollment [Number; unit: participants]
  Japan | 44 | 44 | 41 | 43 | 172
Montgomery Åsberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — MADRS is a10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms.
  units on a scale | 28.5 (5.1) | 28.7 (5.9) | 29.0 (5.4) | 29.3 (5.4) | 28.9 (5.4)
Hamilton Depression Scale 17-Item (HAM D17) [Mean (Standard Deviation); unit: units on a scale] — HAM-D17 is a clinician-rated 17-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 52, where a higher score indicates a greater depressive state.
  units on a scale | 22.6 (2.3) | 22.6 (2.4) | 23.3 (3.0) | 22.9 (2.5) | 22.8 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). Decrease in the total score or on individual items indicates improvement.
Time Frame: Baseline and Week 6
Population: Full Analysis Set: Participants who met the following requirements: major depressive disorder confirmed at registration; at least one dose of the study drug for the treatment period was administered; and at least one efficacy variable was assessed after the start of treatment. Last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Quetiapine 50 mg | Quetiapine 150 mg | Quetiapine 300 mg
Number analyzed (Participants) | 44 | 44 | 41 | 43
units on a scale | -11.5 (1.2) | -11.3 (1.2) | -12.1 (1.2) | -10.3 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Quetiapine 50 mg; Test type: Superiority or Other; Adjusted mean difference = 0.2, 95% CI 2-sided [-3.1 to 3.6], Standard Error of Mean 1.7 — An analysis of covariance model with the baseline as a covariate and treatment group as a fixed effect
Statistical Analysis 2: Comparison: Placebo vs Quetiapine 150 mg; Test type: Superiority or Other; Adjusted mean difference = -0.6, 95% CI 2-sided [-4.0 to 2.8], Standard Error of Mean 1.7 — An analysis of covariance model with the baseline as a covariate and treatment group as a fixed effect
Statistical Analysis 3: Comparison: Placebo vs Quetiapine 300 mg; Test type: Superiority or Other; Adjusted mean difference = 1.3, 95% CI 2-sided [-2.1 to 4.6], Standard Error of Mean 1.7 — An analysis of covariance model with the baseline as a covariate and treatment group as a fixed effect

2. Secondary Outcome: Change From Baseline in Hamilton Rating Score for Depression (HAM-D17)
Description: The 17-item Hamilton Depression Scale (HAM-D17) is a clinician-rated 17-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score range is from 0 to 52 where a higher score indicates a greater depressive state.
Time Frame: Baseline and Week 6
Population: Full analysis set; Last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Quetiapine 50 mg | Quetiapine 150 mg | Quetiapine 300 mg
Number analyzed (Participants) | 44 | 44 | 41 | 43
units on a scale | -10.1 (6.0) | -9.3 (5.9) | -10.2 (5.7) | -8.7 (6.1)

3. Secondary Outcome: Percentage of Participants With Improvement in Clinical Global Impressions-Improvement (CGI-I)
Description: The Clinical Global Impression - global improvement assesses the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale: 1, markedly improved; 2, moderately improved; 3, minimally improved; 4, no change; 5, minimally worsened; 6, moderately worsened; or 7, markedly worsened. Improvement is defined as a score of 1 or 2.
Time Frame: Baseline and Week 6
Population: Full analysis set; Last observation carried forward (LOCF) imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Quetiapine 50 mg | Quetiapine 150 mg | Quetiapine 300 mg
Number analyzed (Participants) | 44 | 44 | 41 | 43
percentage of participants | 54.5 | 50.0 | 53.7 | 27.2

4. Secondary Outcome: Change From Baseline in Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36)
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The 8 health concepts are: 1. Limitation in physical activities because of health problems. 2. Limitations in usual role activities because of physical health problems. 3. Bodily pain. 4. Limitations in social activities because of physical or emotional problems. 5. General mental health (psychological distress and well-being). 6. Limitations in usual role activities because of emotional problems. 7. Vitality (energy and fatigue). 8. General health perception. Each scale ranges from 0 to 100, with 0 indicating the least favorable status and 100 being the most favorable health status.
Time Frame: Baseline and Week 6
Population: Full analysis set with available SF-36 data; LOCF was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Quetiapine 50 mg | Quetiapine 150 mg | Quetiapine 300 mg
Number analyzed (Participants) | 44 | 44 | 39 | 42
units on a scale
  Physical Functioning | 2.8 (13.3) | 1.4 (14.3) | 0.4 (14.9) | 1.4 (12.5)
  Role Limitations - Physical | 8.8 (24.8) | 1.1 (28.0) | 7.4 (31.1) | 6.1 (26.2)
  Bodily pain | 4.4 (21.4) | 11.2 (23.9) | 2.5 (25.2) | -0.5 (26.9)
  General Health Perception | 6.3 (12.3) | 6.0 (14.8) | 4.7 (16.8) | 8.7 (13.5)
  Vitality | 7.5 (15.8) | 8.1 (21.3) | 6.7 (15.8) | 9.2 (18.6)
  Social Functioning | 7.1 (21.3) | 6.5 (27.3) | 7.4 (25.9) | 6.0 (20.3)
  Role Limitations - Emotional | 9.8 (29.5) | 13.8 (24.0) | 11.8 (27.7) | 9.7 (27.3)
  Mental Health | 2.5 (18.9) | 9.7 (22.0) | 8.1 (16.7) | 7.5 (19.4)

5. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction, each on a scale from 0 (best) to 3 (worst). The sum of scores for these seven components yields one global score, ranging from 0 to 21, with higher scores indicative of poor sleep quality.
Time Frame: Baseline and Week 6
Population: Full analysis set with available PSQI data; LOCF was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Quetiapine 50 mg | Quetiapine 150 mg | Quetiapine 300 mg
Number analyzed (Participants) | 44 | 44 | 39 | 42
units on a scale | -1.1 (2.9) | -1.8 (2.7) | -1.5 (2.7) | -1.8 (3.0)

6. Secondary Outcome: Safety Assessed by the Incidence of Adverse Events (AE), Vital Signs, Electrocardiogram (ECG) and Laboratory Tests
Description: An AE is defined as any untoward medical occurrence in a patient administered a study drug, and which does not necessarily have a causal relationship with this treatment. Abnormal laboratory parameters, vital signs or ECG data were defined as AEs if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study medication or was clinically significant. A serious AE was an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, was life-threatening, required or prolonged hospitalization or was considered medically important. AEs were assessed by the Investigator for intensity as mild, moderate or severe and for causal relationship to study drug.
Time Frame: Up to 8 weeks
Measure: Number; unit: participants
Arm/Group | Placebo | Quetiapine 50 mg | Quetiapine 150 mg | Quetiapine 300 mg
Number analyzed (Participants) | 44 | 44 | 41 | 43
participants
  Any adverse event | 25 | 33 | 35 | 35
  Drug-related adverse event | 21 | 24 | 29 | 31
  Deaths | 0 | 0 | 0 | 0
  Serious adverse event | 0 | 1 | 0 | 1
  Drug-related serious adverse event | 0 | 1 | 0 | 1
  AE leading to discontinuation | 2 | 2 | 6 | 4
  Drug-related AE leading to discontinuation | 1 | 2 | 6 | 2

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Placebo | Quetiapine 50 mg | Quetiapine 150 mg | Quetiapine 300 mg
Serious Adverse Events (participants affected / at risk) | 0/44 | 1/44 | 0/41 | 1/43
Other Adverse Events (participants affected / at risk) | 18/44 | 23/44 | 26/41 | 28/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | Quetiapine 50 mg (N=44) | Quetiapine 150 mg (N=41) | Quetiapine 300 mg (N=43)
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | Quetiapine 50 mg (N=44) | Quetiapine 150 mg (N=41) | Quetiapine 300 mg (N=43)
Malaise (General disorders) | 0 | 1 | 1 | 3
Thirst (General disorders) | 2 | 5 | 5 | 9
Nasopharyngitis (Infections and infestations) | 3 | 3 | 6 | 6
Pharyngitis (Infections and infestations) | 3 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 3 | 2
Blood prolactin increased (Investigations) | 3 | 1 | 4 | 2
Blood triglycerides increased (Investigations) | 2 | 6 | 4 | 5
Weight increased (Investigations) | 0 | 2 | 3 | 2
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 6
Dizziness postural (Nervous system disorders) | 1 | 1 | 2 | 4
Headache (Nervous system disorders) | 3 | 5 | 1 | 1
Somnolence (Nervous system disorders) | 6 | 9 | 13 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI needs to get prior approval from Sponsor in writing for publication of trial data.